CLINICAL TRIAL: NCT01881282
Title: A Comparative Clinical Research on Therapeutic Effect and Safety of Compound Carraghenates Cream Versus Mayinglong Musk Hemorrhoid Ointment in the Treatment of Hemorrhoids
Brief Title: A Comparative Efficacy and Safety Study of Compound Carraghenates Cream With Mayinglong Musk Hemorrhoid Ointment in the Treatment of Hemorrhoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002125; TITC-CHN-IIS-02
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Carraghenates; Mayinglong Musk; Titanoreine
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carraghenates Cream (Experimental)
  Interventions: Drug: Carraghenates Cream
- Mayinglong Musk Hemorrhoid Ointment (Active Comparator)
  Interventions: Drug: Mayinglong Musk Hemorrhoid Ointment

INTERVENTIONS:
Drug: Carraghenates Cream — Carraghenates cream will be administered 3-4 gram (g) each time (one sixth of a piece) through anal canal, twice a day (once in the morning and once in the evening); for consecutive 6 days.
  Arms: Carraghenates Cream
Drug: Mayinglong Musk Hemorrhoid Ointment — Mayinglong musk hemorrhoid ointment will be administered 2 g each time through anal canal, twice a day (once in the morning and once in the evening) for consecutive 6 days.
  Arms: Mayinglong Musk Hemorrhoid Ointment

SUMMARY:
The purpose of this study is to compare the therapeutic effect and safety of compound carraghenates cream with Mayinglong musk hemorrhoid (swollen veins in the lower part of the rectum or anus) ointment in the treatment of hemorrhoids, especially regarding the relief of pain.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (study drug assigned by chance), multi-center (when more than one hospital or medical school team work on a medical research study), controlled clinical trial and comparative study of safety and efficacy of compound carraghenates cream with Mayinglong musk hemorrhoid ointment in the treatment of hemorrhoids, especially regarding the relief of pain. Participants will be randomly assigned to either of the two treatment groups that are carraghenates cream (Titanoreine) group or Mayinglong musk hemorrhoid ointment group. The total duration of the study will be 1 Week (7 days). In carraghenates cream group, 3-4 gram (g) cream will be administered each time through anal canal, twice a day, once in the morning and once in the evening for consecutive 6 days and in the Mayinglong musk hemorrhoid ointment group, 2 g ointment will be administered each time through anal canal, twice a day, once in the morning and once in the evening for consecutive 6 days. Efficacy will be assessed by using Numeric Rating Scale (NRS) and participants' safety will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants who agree to participate in the current study
* Participants having painful hemorrhoids (swollen veins in the lower part of the rectum or anus [external hemorrhoid, mixed hemorrhoid, etc.])
* Participants who did not use other topical drugs to treat their hemorrhoids a day before the inclusion
* Participants who do not use drugs other than the study drug and the control drug to treat their hemorrhoids during the study period

Exclusion Criteria:

* Participants having other anorectal diseases , such as anal fistula , anal cleft , perianal abscess , and anorectal occupied lesions etc
* Participants having hypersensitive predisposition or hypersensitive to any of components of the study drugs
* Female participants under pregnancy or during breastfeeding period
* Participants who fail to accept the scheduled visits or are lost to the visits
* Participants complicated by serious cardio cerebro vascular diseases, hepatic and renal diseases, diseases of hemopoietic system or mental disorders

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pain Acting Time | Day 1 up to Day 7
  The time from the first administration of the drugs to the time when the participant feels that his (her) pain has been remitted remarkably will be assessed.
Pain Intensity Score at Day 4 | Day 4
  Pain intensity will be measured on an 11-point numeric rating scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates intense pain. Grade 1-4 represents mild pain, Grade 5-6 moderate pain, and Grade 7-10 serious pain. Higher score indicates worsening.
Pain Intensity Score at Day 7 | Day 7
  Pain intensity will be measured on an 11-point numeric rating scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates intense pain. Grade 1-4 represents mild pain, Grade 5-6 moderate pain, and Grade 7-10 serious pain. Higher score indicates worsening.
Daily Duration of Symptoms | Day 1 up to Day 7
  The accumulated time of the onset of all symptoms in the same day will be assessed. The baseline value before the administration of the drugs is the accumulated time of the occurrence of all symptoms in the day prior to the visit.
Frequency of Defecation | Day 1 up to Day 7
  The daily frequency of defecation for the day prior to the visit and each day during the trial period will be assessed.
Participants' Satisfaction for the Treatment | Day 7
  Participants' will assess for the treatment satisfaction on numeric rating scale (NRS) ranging from 1 to 5, where 1= Very unsatisfactory; 2= Unsatisfactory; 3=General; 4= Satisfactory; 5= Very satisfactory.
Assessment of Other Symptoms and Signs Including Bleeding, Edema, Local Discomfort, and Prolapse | Day 1 up to Day 7
  Participants will assess these symptoms on a score range of 0 to 3 where 0=none for all symptoms and 3= "Blood jets while defecating, and the blood jetting stops after defecation" for bleeding, "serious edema" for edema, "severe" for local discomfort and "it is difficult or unable to return the prolapsed pile" for prolapse.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development LLC Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.